CLINICAL TRIAL: NCT01221610
Title: A Prospective, Multi-centre, Randomized Controlled, First in Man Study to Assess the Safety and Performance of the Passeo-18 Lux Paclitaxel Releasing PTA Balloon Catheter vs. the Uncoated Passeo 18 Balloon Catheter in Patients With Stenosis and Occlusion of the Femoropopliteal Arteries (BIOLUX P-I).
Brief Title: BIOLUX P-I First in Man Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1003
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Atherosclerosis; Arteriosclerosis; Vascular Disease; Peripheral Artery Disease
Keywords: Stenosis; Occlusions; SFA; PTA; POBA; DRB
MeSH Terms: conditions — Atherosclerosis; Arteriosclerosis; Vascular Diseases; Peripheral Arterial Disease; Constriction, Pathologic; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug Releasing Balloon (Experimental): Passeo-18 Lux Drug Releasing Balloon catheter
  Interventions: Device: Passeo-18 Lux DRB
- Standard PT A (POBA) (Active Comparator): Uncoated Passeo-18 PTA catheter
  Interventions: Device: Standard PTA (POBA)

INTERVENTIONS:
Device: Passeo-18 Lux DRB
  Other Names: Passeo-18 Lux Drug Releasing Balloon catheter
  Arms: Drug Releasing Balloon
Device: Standard PTA (POBA)
  Other Names: Passeo-18 PTA catheter
  Arms: Standard PT A (POBA)

SUMMARY:
A prospective, multi-centre, randomized controlled, First in Man study to assess the safety and performance of the coated Passeo-18 Lux Paclitaxel releasing PTA Balloon Catheter vs. an uncoated balloon catheter in patients with stenosis and occlusion of the femoropopliteal arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years,
2. Informed consent signed by patient prior to randomization
3. Single or sequential de novo or restenotic lesions (stenosis ≥ 70% diameter reduction or occlusion) in the femoropopliteal arteries ≥ 30 mm and ≤ 200 mm long
4. Rutherford Class 2 - 5 in the target limb
5. Reference Vessel Diameter (RVD) 3 - 7 mm, based on visual estimation
6. Inflow free from flow-limiting lesion (< 50% stenosis) confirmed by angiography. Patients with flow-limiting inflow lesions (> 50% stenosis) can be included if lesion has been treated successfully before the index procedure
7. At least one non-occluded crural vessel (eg without significant stenosis) with angiographically documented run-off to the foot
8. Successful wire crossing of the lesion
9. Willingness to comply with all specified follow-up evaluations
10. Male or negative pregnancy test of women in childbearing age

Exclusion Criteria:

1. Co-morbid conditions limiting life expectancy ≤ 1 year
2. Patient currently participating in another clinical trial
3. Lesions which are untreatable with PTA or other interventional techniques
4. The target stenosis is located distal to a stenosis ≥ 50% that cannot be pre-treated because the drug coating could get lost during crossing the proximal lesion
5. Thrombus in the target vessel, documented by angiography
6. Target lesion is severely calcified, documented by angiography
7. Prior bypass surgery of target vessel
8. Previously implanted stent in the target lesion
9. Treatment of bifurcation required
10. Planned amputation of the target limb
11. Flow-limiting (> 50% DS) Inflow lesion proximal to target lesion, left untreated
12. Failure to obtain <30% residual stenosis in a pre-existing haemodynamically significant (>50% DS) inflow lesion in the ipsilateral iliac or proximal SFA. (DEB or DES not allowed for the treatment of inflow lesion)
13. Additional hemodynamically relevant proximal and distal lesions with stenosis ≥ 50 %, except iliac arteries, are excluded. Iliac artery lesion treatments have to be successful with a residual stenosis ≤ 30 %
14. Haemorrhagic diathesis or another disorder such as gastrointestinal ulceration or cerebral circulatory disorders which restrict the use of platelet aggregation inhibitor therapy and anticoagulation therapy
15. Phenprocoumon intake
16. Impaired renal function (creatinine ≥ 2.0 - 2.5 mg/dl), according to investigator assessment
17. Known allergy to contrast media that cannot be adequately controlled with pre-medication
18. Allergy, intolerance or hypersensitivity to Paclitaxel structurally or related compounds and/or to the delivery matrix n-Butyryl tri-nhexyl citrate (BTHC)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-10; Primary Completion 2012-02 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the 6 months late lumen loss in the target lesion measured by quantitative vascular angiography (QVA). | 6 months

SECONDARY OUTCOMES:
6 months binary restenosis rate | 6 months
6 months and 12 months TLR rate | 6 and 12 months
6 months and 12 months change in mean ABI | 6 and 12 months
6 months and 12 months change in Rutherford class | 6 and 12 months
Major Adverse Event rate at 6 and 12 months (procedure- or device-related death or amputation, target lesion thrombosis and clinically driven TLR) | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, MD, Principal Investigator — Park-Krankenhaus Leipzig GmbH, Leipzig, Germany
Locations (5):
- AKH Wien, Kardiovaskuläre und Interventionelle Radiologie, Vienna, Austria
- Germany (4):
  - Universitäts-Herzzentrum Freiburg Bad Krozingen, Bad Krozingen
  - Gefaesszentrum Berlin, Medizinische Klinik, Ev. Krankenhaus Königin Elisabeth Herzberge, Berlin
  - Parkkrankenhaus Leipzig Südost GmbH, Leipzig
  - Institut für diagnostische und interventionelle Radiologie, Klinikum Rosenheim, Rosenheim